CLINICAL TRIAL: NCT02545933
Title: Adjunctive Vorapaxar Therapy in Patients With Prior Myocardial Infarction Treated With New Generation P2Y12 Receptor Inhibitors Prasugrel and Ticagrelor (VORA-PRATIC): A Prospective, Randomized, Pharmacodynamic Study
Brief Title: Vorapaxar in Patients With Prior Myocardial Infarction Treated With Prasugrel and Ticagrelor
Acronym: VORA-PRATIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS 53376
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Myocardial Infarction
Keywords: prasugrel; ticagrelor; vorapaxar
MeSH Terms: conditions — Myocardial Infarction | interventions — Prasugrel Hydrochloride; vorapaxar; Aspirin; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DAPT plus vorapaxar (Experimental): Aspirin plus prasugrel or ticagrelor plus vorapaxar 2.5mg od
  Interventions: Drug: Prasugrel; Drug: Vorapaxar; Drug: Aspirin; Drug: Ticagrelor
- Prasugrel/ticagrelor plus vorapaxar (Experimental): Prasugrel or ticagrelor plus vorapaxar 2.5mg od
  Interventions: Drug: Prasugrel; Drug: Vorapaxar; Drug: Ticagrelor
- DAPT (Active Comparator): Aspirin in addition to prasugrel or ticagrelor
  Interventions: Drug: Prasugrel; Drug: Aspirin; Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Patients will continue treatment with either prasugrel (10mg once daily) or ticagrelor (90mg twice/daily)
  Other Names: Effient
Drug: Vorapaxar — Vorapaxar will be administered at the dose of 2.5mg once daily
  Other Names: Zontivity
  Arms: DAPT plus vorapaxar; Prasugrel/ticagrelor plus vorapaxar
Drug: Aspirin — Aspirin will be administered at the dose of 81mg once daily
  Other Names: ASA (acetylsalicylic acid)
  Arms: DAPT; DAPT plus vorapaxar
Drug: Ticagrelor — Patients will continue treatment with either prasugrel (10mg once daily) or ticagrelor (90mg twice/daily)
  Other Names: Brilinta

SUMMARY:
Dual antiplatelet therapy (DAPT) with aspirin and a P2Y12 receptor inhibitor represents the standard of care for the long-term secondary prevention of atherothrombotic events in patients with myocardial infarction (MI). However, rates of ischemic recurrences remain high, which may be in part due to the fact that other platelet signaling pathways, such as thrombin-induced platelet aggregation, continue to be activated. Vorapaxar is a protease-activated receptor (PAR)-1 inhibitor, which exerts potent inhibition of thrombin-mediated platelet aggregation. It is approved for clinical use by the Food and Drug Administration for the reduction of thrombotic cardiovascular events in patients with a history of MI or with peripheral arterial disease. However, to date clinical trial experience with vorapaxar has been almost exclusively with the P2Y12 receptor inhibitor clopidogrel and the effects of vorapaxar in combination with antiplatelet therapy including prasugrel or ticagrelor, is largely unexplored. Further, the role of vorapaxar as part of a dual antithrombotic treatment regimen, in addition to a novel P2Y12 receptor inhibitor, with withdrawal of aspirin, represents another important area of clinical interest as it has the potential to maximize ischemic protection while reducing the risk of bleeding. The proposed prospective, randomized, parallel-design, open label, study conducted in a real world clinical setting of post-MI patients will aim to assess the pharmacodynamic effects of vorapaxar in addition to antiplatelet therapy with a novel P2Y12 receptor inhibitor (prasugrel or ticagrelor) with and without aspirin.

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) with aspirin and a P2Y12 receptor inhibitor represents the standard of care for the long-term secondary prevention of atherothrombotic events in patients with myocardial infarction (MI). The novel P2Y12 receptor inhibitors prasugrel and ticagrelor are characterized by more prompt, potent, and predictable antiplatelet effects compared with clopidogrel and are associated with a greater reduction of ischemic events in acute coronary syndrome patients. However, rates of ischemic recurrences remain high, which may be in part due to the fact that other platelet signaling pathways, such as thrombin-induced platelet aggregation, continue to be activated. Vorapaxar is a novel, orally active, competitive and slowly reversible protease-activated receptor (PAR)-1 inhibitor, which exerts potent inhibition of thrombin-mediated platelet aggregation. It is approved for clinical use by the Food and Drug Administration for the reduction of thrombotic cardiovascular events in patients with a history of MI or with peripheral arterial disease. A large-scale clinical trial showed that the use of vorapaxar (2.5 mg once/daily) in addition to standard antiplatelet therapy (including aspirin and a P2Y12 receptor inhibitor) was effective in the secondary prevention of recurrent thrombotic events in patients with previous atherothrombosis, in particular in patients with prior MI, at the expense of an increase in major bleeding. However, to date clinical trial experience with vorapaxar has been almost exclusively with the P2Y12 receptor inhibitor clopidogrel and the effects of vorapaxar in combination with state-of-the-art antiplatelet therapy in the post-MI setting, including prasugrel or ticagrelor, is largely unexplored. This may indeed represent a limitation for the uptake of vorapaxar in modern day clinical practice where these agents are being more broadly utilized. Further, the role of vorapaxar as part of a dual antithrombotic treatment regimen, in addition to a novel P2Y12 receptor inhibitor, with withdrawal of aspirin, represents another important area of clinical interest as it has the potential to maximize ischemic protection while reducing the risk of bleeding. The proposed prospective, randomized, parallel-design, open label, study conducted in a real world clinical setting of post-MI patients will aim to assess the pharmacodynamic effects of vorapaxar in addition to antiplatelet therapy with a novel P2Y12 receptor inhibitor (prasugrel or ticagrelor) with and without aspirin. Pharmacodynamic assessments will be performed at multiple time points and with different assays exploring multiple pathways of platelet aggregation. Exploratory assessments on the safety of such approach will also be evaluated.

ELIGIBILITY:
Inclusion criteria:

1. Patients with a prior MI within the previous 2 weeks to 12 months.
2. On DAPT with low-dose aspirin (81mg od) and either prasugrel (10mg od) or ticagrelor (90mg bid) as per standard-of-care for at least 2 weeks.
3. Free from bleeding and ischemic events after the index MI event.
4. Age between 18 and 75 years old.

Exclusion criteria:

1. History of stroke, transient ischemic attack, or intracranial hemorrhage.
2. Active pathological bleeding, history of bleeding events or increased risk of bleeding.
3. Known severe hepatic impairment.
4. Age >75 years.
5. Body weight <60 Kg.
6. Use of strong Cytochrome P450 3A inhibitors (e.g., ketoconazole, itraconazole, posaconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, boceprevir, telaprevir, telithromycin and conivaptan) or inducers (e.g., rifampin, carbamazepine, St. John's Wort and phenytoin).
7. On treatment with any oral anticoagulant (vitamin K antagonists, dabigatran, rivaroxaban, apixaban, edoxaban).
8. On treatment with any antiplatelet agent other than aspirin, prasugrel and ticagrelor in the past 14 days.
9. Creatinine clearance <30 mL/minute.
10. Platelet count <80x106/mL
11. Hemoglobin <10g/dL
12. Hemodynamic instability
13. Pregnant females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD, PhD, Principal Investigator — University of Florida College of Medicine-Jacksonville
Locations (1):
- University of Florida, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Franchi F, Rollini F, Faz G, Rivas JR, Rivas A, Agarwal M, Briceno M, Wali M, Nawaz A, Silva G, Shaikh Z, Maaliki N, Fahmi K, Been L, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Baber U, Mehran R, Jennings LK, Bass TA, Angiolillo DJ. Pharmacodynamic Effects of Vorapaxar in Prior Myocardial Infarction Patients Treated With Potent Oral P2Y12 Receptor Inhibitors With and Without Aspirin: Results of the VORA-PRATIC Study. J Am Heart Assoc. 2020 Apr 21;9(8):e015865. doi: 10.1161/JAHA.120.015865. Epub 2020 Apr 20. PMID 32306797

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DAPT Plus Vorapaxar | Prasugrel/Ticagrelor Plus Vorapaxar | DAPT
Started | 44 | 43 | 43
Completed | 38 | 40 | 39
Not Completed | 6 | 3 | 4
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 3
Not completed — Protocol Violation | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DAPT Plus Vorapaxar | Prasugrel/Ticagrelor Plus Vorapaxar | DAPT | Total
Number analyzed (Participants) | 44 | 43 | 43 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9) | 56 (9) | 56 (10) | 56 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 14 | 39
  Male | 30 | 32 | 29 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 14 | 13 | 44
  White | 24 | 26 | 29 | 79
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44 | 43 | 43 | 130
Diabetes mellitus [Count of Participants; unit: Participants] | 11 | 12 | 10 | 33

OUTCOME MEASURES:

1. Primary Outcome: Maximal Platelet Aggregation
Description: The primary end point of our study is the comparison of maximal platelet aggregation measured by light transmittance aggregometry using CAT (collagen-ADP-TRAP) between DAPT and DAPT plus vorapaxar after 30 days of treatment.
Time Frame: 30 days
Population: 130 patients were randomized and exposed to at least one dose of study medication (triple therapy, n=44; dual therapy, n= 43; DAPT, n=43). Of these, 115 patients (triple therapy, n=37; dual therapy, n= 39; DAPT, n=39) had valid primary endpoint data
Measure: Mean (Standard Deviation); unit: percent aggregation
Arm/Group | DAPT Plus Vorapaxar | Prasugrel/Ticagrelor Plus Vorapaxar | DAPT
Number analyzed (Participants) | 37 | 39 | 39
percent aggregation | 52 (21) | 64 (20) | 74 (10)
Statistical Analysis 1: Comparison: DAPT Plus Vorapaxar vs Prasugrel/Ticagrelor Plus Vorapaxar vs DAPT; We hypothesized that adjunctive vorapaxar would result in a significant reduction of CAT-induced platelet aggregation. Assuming a 10% absolute reduction in CAT-induced maximal platelet aggregation with a common standard deviation of 13%, 37 patients per group with valid primary endpoint data were required to detect a significant difference with a 90% power and 2-sided alpha=0.05; Test type: Superiority; p = 0.011, ANOVA; least square mean difference = 27, 95% CI 2-sided [19 to 34] — DAPT group vs DAPT plus vorapaxar group

ADVERSE EVENTS:
Time Frame: Duration of the study (30 days)
Arm/Group | DAPT Plus Vorapaxar | Prasugrel/Ticagrelor Plus Vorapaxar | DAPT
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 9/44 | 6/43 | 4/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DAPT Plus Vorapaxar (N=44) | Prasugrel/Ticagrelor Plus Vorapaxar (N=43) | DAPT (N=43)
BARC 1 bleeding (Blood and lymphatic system disorders) | 6 (6) | 1 (1) | 0 (0) — BARC (Bleeding Academic Research Consortium) 1 bleeding
chest pain (Cardiac disorders) | 0 | 0 | 4
diarrhea (Gastrointestinal disorders) | 1 | 2 | 0
dizziness (General disorders) | 1 | 2 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-06-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT02545933/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT02545933/ICF_001.pdf